CLINICAL TRIAL: NCT06418997
Title: Cognitive Behavioral Immersion: A Randomized Control Trial of Peer-Based Coaching in the Metaverse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Iony Ezawa, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UP-23-00491; R44MH132202 (NIH)
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-01

CONDITIONS: Depression, Anxiety
Keywords: Metaverse; virtual reality; cognitive-behavioral; depression; depressive Disorders; mental disorders; skills group
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBI-Virtual Reality (Active Comparator): Over 8 weekly 1-hour sessions, participants will learn about the cognitive-behavioral model from trained peer coaches, develop cognitive-behavioral skills that they can utilize in their daily lives (such as cognitive restructuring), and engage with a receptive community of peers. Participants randomized to this arm will access these sessions using a virtual reality headset.
  Interventions: Behavioral: CBI
- CBI-Flat Screen (Active Comparator): Over 8 weekly 1-hour sessions, participants will learn about the cognitive-behavioral model from trained peer coaches, develop cognitive-behavioral skills and habits that they can utilize in their daily lives (such as cognitive restructuring), and engage with a receptive community of peers. Participants randomized to this arm will access these sessions using a flat-screen device, such as a computer.
  Interventions: Behavioral: CBI
- Delayed-Access Control (No Intervention): Participants randomized to this arm will be asked not to attend CBI sessions.

INTERVENTIONS:
Behavioral: CBI — CBI sessions follow a detailed manual to teach a group of peers cognitive and behavioral strategies that they may utilize in their daily lives, often based around the cognitive-behavioral model as a teaching tool. CBI aims to develop cognitive-behaviorally-based skills and habits in participants, such as behavioral activation, mood tracking, the identification and reframing of automatic thoughts, and assertion training.
  Arms: CBI-Flat Screen; CBI-Virtual Reality

SUMMARY:
This study will test a new cognitive-behavioral skills training program (CBI) delivered in the metaverse. Although initial evidence suggested CBI was feasible for individuals experiencing depression or anxiety, CBI's effectiveness compared to no intervention has yet to be determined. The intervention may be delivered through virtual reality as well as flat-screen devices, such as a computer, which may also affect CBI's effectiveness.

The study will enroll up to 306 participants with depression. One third of the participants will access CBI through virtual reality, one third of the participants will access CBI through a flat-screen device, and one third of the participants will be asked not to attend CBI sessions for the first 8 weeks of participation of the trial. For both CBI conditions, treatment will be provided over 8 weeks, with a 6-month follow-up period. Enrollment will be ongoing and groups will occur simultaneously.

Potential participants are asked to complete an initial screening and an intake evaluation to determine eligibility. They will then receive 8-weeks of treatment. Participants will complete brief weekly self-report questionnaires throughout their time in the study.

DETAILED DESCRIPTION:
Cognitive behavioral therapy (CBT) is one of the most effective tools for the treatment of depression and anxiety. Despite its many strengths, CBT-based clinical care is often very expensive and difficult to access. To address problems of accessibility, the field is increasingly utilizing lay therapists (also commonly referred to as coaches or peers) to provide cognitive behavioral coaching. There is also accumulating evidence indicating that technology can be used to deliver affordable and accessible treatments with outcomes comparable to traditional face-to-face psychotherapy treatments (Karyotaki et al., 2021). In particular, the metaverse (Internet-connected 3-D virtual environments have also that allow end-users to interact as avatars) may be a distinctively powerful medium through which to deliver engaging, affordable, accessible, and scalable mental health interventions. In addition, the use of social virtual reality (VR) mental health interventions is relatively unexplored, yet the sense of presence ("being there") it provides may be useful to increase immersiveness in a digital intervention or facilitate social interaction in a digital space.

Therefore, the investigators plan to conduct a randomized controlled trial on CBI in order to investigate its effectiveness among different groups of people and investigate the role immersive VR, as opposed to a flat screen, may play in predicting outcome measures. Upon joining the study, participants are asked to complete surveys once a week for 8 weeks and brief monthly follow-up surveys for 6 months. If you are randomized to either of the CBI conditions, you will also be asked to attend 8 weekly 1-hour sessions through a virtual application (from a VR headset or flat-screen, depending on your condition). This study seeks to address the main following research questions: (1) Is CBI efficacious? (and for whom is it more or less efficacious?) And (2) Does immersive VR confer any advantage over and above accessing CBI via less immersive flat screen devices?

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Proficient in reading and speaking English
* Have a computer with a stable internet connection
* Score at or above the clinical threshold on the Patient Health Questionnaire (PHQ-9; Kroenke et al. 2001)

Exclusion Criteria:

* Sufficiently elevated levels of negative thoughts such that the individual is considered at high risk of harm, according to the Columbia Suicide Severity Rating Scale (CSSRS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Post-treatment (8-weeks) and follow-up (6-months)
  The PHQ-9 (Kroenke et al., 2001) is a 9-item self-report measure with strong psychometric properties that mirrors the nine criteria for evaluating whether someone meets criteria for major depressive disorder (MDD) in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV; American Psychiatric Association, 1994). Scores range from 0 to 27, with higher scores indicating great symptom severity.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Questionnaire (GAD-7) | Post-treatment (8-weeks) and follow-up (6-months)
  The GAD-7 (Spitzer et al., 2006) is a 7-item self-report measure with strong psychometric properties based on the diagnostic criteria for Generalized Anxiety Disorder (GAD-7) from the DSM-IV (American Psychiatric Association, 1994). Scores range from 0 to 21, with higher scores indicating great symptom severity.
WHO Quality of Life-Brief (QOL) | Post-treatment (8-weeks) and 1-item version at follow-up (6-months)
  The WHO QOL (Whoqol Group, 1998) is a 26-item self-report cross-cultural measure of quality of life within the domains of physical health, psychological health, social relationships, and environment. During the follow-up period, we will transition to using only the first item of the measure assessing overall quality of life. Scores are transformed on a scale from 0 to 100, with higher scores indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Iony D Ezawa, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karyotaki E, Efthimiou O, Miguel C, Bermpohl FMG, Furukawa TA, Cuijpers P; Individual Patient Data Meta-Analyses for Depression (IPDMA-DE) Collaboration; Riper H, Patel V, Mira A, Gemmil AW, Yeung AS, Lange A, Williams AD, Mackinnon A, Geraedts A, van Straten A, Meyer B, Bjorkelund C, Knaevelsrud C, Beevers CG, Botella C, Strunk DR, Mohr DC, Ebert DD, Kessler D, Richards D, Littlewood E, Forsell E, Feng F, Wang F, Andersson G, Hadjistavropoulos H, Christensen H, Ezawa ID, Choi I, Rosso IM, Klein JP, Shumake J, Garcia-Campayo J, Milgrom J, Smith J, Montero-Marin J, Newby JM, Breton-Lopez J, Schneider J, Vernmark K, Bucker L, Sheeber LB, Warmerdam L, Farrer L, Heinrich M, Huibers MJH, Kivi M, Kraepelien M, Forand NR, Pugh N, Lindefors N, Lintvedt O, Zagorscak P, Carlbring P, Phillips R, Johansson R, Kessler RC, Brabyn S, Perini S, Rauch SL, Gilbody S, Moritz S, Berger T, Pop V, Kaldo V, Spek V, Forsell Y. Internet-Based Cognitive Behavioral Therapy for Depression: A Systematic Review and Individual Patient Data Network Meta-analysis. JAMA Psychiatry. 2021 Apr 1;78(4):361-371. doi: 10.1001/jamapsychiatry.2020.4364. PMID 33471111
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Derived] Robinson N, Ramos FN, Hollon SD, Han GT, Ezawa ID. Cognitive Behavioral Immersion for Depression: Protocol for a Three-Arm Randomized Controlled Trial of Peer-Based Coaching in the Metaverse. JMIR Res Protoc. 2025 May 6;14:e65970. doi: 10.2196/65970. PMID 40327374